CLINICAL TRIAL: NCT01426412
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3015014 in Subjects With Elevated LDL-C
Brief Title: A Study of LY3015014 in Healthy Participants With Elevated Low Density Lipoprotein Cholesterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13980; I5S-EW-EFJA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY3015014 intravenously (IV) (Experimental): A single dose of LY3015014 up to 10.0 milligrams per kilogram (mg/kg) administered IV
  Interventions: Drug: LY3015014 IV
- LY3015014 IV Japanese (Experimental): Single dose of LY3015014 10.0 mg/kg administered IV to Japanese participants. Added per protocol amendment effective October, 2012.
  Interventions: Drug: LY3015014 IV
- Placebo IV (Placebo Comparator): Administered IV once only
  Interventions: Drug: Placebo IV
- LY3015014 subcutaneously (SC) (Experimental): A single dose of LY3015014 up to 3.0 mg/kg administered SC
  Interventions: Drug: LY3015014 SC
- LY3015014 SC + Statin (Experimental): A single dose of LY3015014 up to 3 mg/kg administered SC in addition to participant's dose of statin
  Interventions: Drug: LY3015014 SC
- Placebo SC (Placebo Comparator): Administered SC once only
  Interventions: Drug: Placebo SC

INTERVENTIONS:
Drug: LY3015014 IV — Administered IV over 30-90 minutes
  Arms: LY3015014 IV Japanese; LY3015014 intravenously (IV)
Drug: Placebo IV — Administered IV only over 30-90 minutes
  Arms: Placebo IV
Drug: LY3015014 SC — Administered SC
  Arms: LY3015014 SC + Statin; LY3015014 subcutaneously (SC)
Drug: Placebo SC — Administered SC
  Arms: Placebo SC

SUMMARY:
This is a study in otherwise healthy Japanese and non-Japanese participants with elevated low density lipoprotein cholesterol (LDL-C). Following single doses of LY3015014, the safety and tolerability of the drug, how the body handles the drug, and the drug's effect on the body will be evaluated. Participants will remain in the study for approximately up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* To qualify as Japanese for the purpose of this study, the participant must be first-generation Japanese, defined as the participant's biological parents and all of the participant's biological grandparents must be of exclusive Japanese descent, and must have been born in Japan. Japanese participants have to be between the ages of 20-65, inclusive, at screening
* Statin naive participants, have a screening LDL-C of between 100 and 180 milligrams per deciliter (mg/dL), inclusive; for participants currently taking a statin, have a screening LDL-C of between 100 and 160 mg/dL
* Have serum triglycerides <400 mg/dL

Additional inclusion criteria for participants in the statin-interaction cohort:

* At screening, must have been on a stable dose of either atorvastatin [10 to 40 mg once daily (QD)], rosuvastatin (5 to 20 mg QD), simvastatin (20 to 40 mg QD), lovastatin (40 to 80 mg QD), or pravastatin (40 to 80 mg QD) which has been well tolerated for at least 3 months

Exclusion Criteria:

* Have known allergies to compounds related to LY3015014 or any components of the formulation, or known clinically significant hypersensitivity to biologic agents, or known allergies to acetaminophen and/or antihistamines
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing (excluding the statins listed in Inclusion Criterion), other than estrogen/progesterone as hormone replacement therapy (HRT) and thyroid medications. Participants taking these medications should be on chronic, stable doses. Certain medications, for example vitamin supplements, may be permitted at the discretion of the investigator and the sponsor. Participants on statins may be allowed to be on a stable dose of single hypertensive agent if agreed upon by sponsor and investigator
* Have received any vaccine(s) within 1 month of LY3015014 dosing, or intend to during the study
* Have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Have a history of atopy, or significant allergies to humanized monoclonal antibodies, or clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions [including, but not limited to, erythema multiforme major, linear immunoglobulin (Ig)A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis]

Additional exclusion criteria for participants in the statin-interaction cohort:

* Incidence of unexplained muscle pain, or incidence of frequent muscle cramp within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.03 mg/kg LY3015014 IV: A single dose of 0.03 milligrams per kilogram (mg/kg) LY3015014 administered intravenously (IV).
- 0.1 mg/kg LY3015014 IV: A single dose of 0.1 mg/kg LY3015014 administered IV.
- 0.3 mg/kg LY3015014 IV: A single dose of 0.3 mg/kg LY3015014 administered IV.
- 1.0 mg/kg LY3015014 IV: A single dose of 1.0 mg/kg LY3015014 administered IV.
- 3.0 mg/kg LY3015014 IV: A single dose of 3.0 mg/kg LY3015014 administered IV.
- 3.0 mg/kg LY3015014 SC: A single dose of 3.0 mg/kg LY3015014 administered SC.
- 3.0 mg/kg LY3015014 SC +Statin: A single dose of 3.0 mg/kg LY3015014 administered subcutaneously (SC) with a statin add-on dose.
- 10.0 mg/kg LY3015014 IV: A single dose of 10.0 mg/kg LY3015014 administered IV to non-Japanese or Japanese participants.
- Placebo: A single dose of placebo administered IV or SC with a statin add-on dose.
Period: Overall Study
Arm/Group | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin | 10.0 mg/kg LY3015014 IV | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 17
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 17
Completed | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 7 | 16
Not Completed | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin | 10.0 mg/kg LY3015014 IV | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 17 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (8.6) | 47.3 (10.3) | 46.3 (17.5) | 50.2 (14.6) | 51.7 (13.9) | 44.3 (14.1) | 53.3 (4.1) | 52.5 (12.0) | 48.5 (12.8) | 49.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 2 | 2 | 1 | 4 | 7 | 23
  Male | 5 | 4 | 4 | 4 | 4 | 4 | 5 | 6 | 10 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 6
  Not Hispanic or Latino | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 8 | 16 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 7
  White | 5 | 6 | 6 | 6 | 6 | 5 | 4 | 4 | 14 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Adverse events (AEs) were considered as clinically significant effects. A summary of serious AEs (SAEs) and other nonserious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion (up to 22 weeks)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- 0.03 mg/kg LY3015014 IV: A single dose of 0.03 mg/kg LY3015014 administered IV.
- 3.0 mg/kg LY3015014 SC +Statin: A single dose of 3.0 mg/kg LY3015014 administered SC with a statin add-on dose.
Arm/Group | Placebo | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin | 10.0 mg/kg LY3015014 IV
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE | 13 | 4 | 4 | 2 | 3 | 3 | 6 | 3 | 6

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Time 0 to the Last Time Point With a Measurable Concentration of LY3015014 [AUC(0-tlast)]
Time Frame: Predose, 0, 1, 2, 4, 12, 24 hours post dose, and 3, 5, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 85, 99, 113, 127 and 155 days post-dose
Population: All randomized participants who received LY3015014 and had PK data to calculate AUC(0-tlast).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms *hour/milliliter (µg*h/mL)
Groups:
- 10.0 mg/kg LY3015014 IV Non-Japanese: A single dose of 10.0 mg/kg LY3015014 administered IV to non-Japanese participants.
- 10.0 mg/kg LY3015014 IV Japanese: A single dose of 10.0 mg/kg LY3015014 administered IV to Japanese participants.
Arm/Group | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 10.0 mg/kg LY3015014 IV Non-Japanese | 10.0 mg/kg LY3015014 IV Japanese | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 6 | 4 | 6 | 6
micrograms *hour/milliliter (µg*h/mL) | 109 (9) | 435 (16) | 1450 (20) | 5610 (22) | 18600 (17) | 89100 (17) | 57500 (62) | 12700 (39) | 11700 (32)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3015014
Time Frame: as for outcome 2
Population: All randomized participants who received LY3015014 and had PK data to calculate Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 10.0 mg/kg LY3015014 IV Non-Japanese | 10.0 mg/kg LY3015014 IV Japanese | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 6 | 4 | 6 | 6
micrograms per milliliter (µg/mL) | 1.18 (16) | 3.18 (7) | 11.0 (18) | 29.2 (21) | 97.3 (27) | 312 (18) | 282 (9) | 24.8 (25) | 19.8 (24)

4. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Least Square means were calculated using mixed-effects models for repeated measures analysis. The model included factors for treatment, visits and baseline LDL-C. Percent change = (LDL value on Days 15 or 29 - LDL at baseline) / LDL at baseline *100.
Time Frame: Baseline, Days 15 and 29
Population: All randomized participants with evaluable LDL-C data at specified time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of change
Arm/Group | Placebo | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin | 10.0 mg/kg LY3015014 IV Japanese | 10.0 mg/kg LY3015014 IV Non-Japanese
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 6
percentage of change
  Day 15 | -1.69 [-6.56 to 3.19] | -11.55 [-19.79 to -3.32] | -17.49 [-25.70 to -9.27] | -40.34 [-48.56 to -32.12] | -34.84 [-43.08 to -26.59] | -57.00 [-65.21 to -48.79] | -53.56 [-61.78 to -45.34] | -56.58 [-64.83 to -48.33] | -47.31 [-58.35 to -36.28] | -50.83 [-59.03 to -42.62]
  Day 29 | -2.88 [-7.75 to 2.00] | -6.17 [-14.89 to 2.55] | -13.01 [-21.22 to -4.80] | -31.83 [-40.05 to -23.60] | -34.90 [-43.15 to -26.65] | -54.40 [-62.61 to -46.19] | -51.63 [-59.85 to -43.40] | -58.02 [-66.27 to -49.76] | -39.31 [-52.51 to -26.10] | -58.08 [-66.28 to -49.87]

5. Secondary Outcome: Number of Participants With Detectable Levels of Anti-LY3015014 Antibodies
Time Frame: Days 8, 29 and 85
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin | 10.0 mg/kg LY3015014 IV
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Day 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up To 22 weeks
Arm/Group | 0.03 mg/kg LY3015014 IV | 0.1 mg/kg LY3015014 IV | 0.3 mg/kg LY3015014 IV | 1.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 IV | 3.0 mg/kg LY3015014 SC | 3.0 mg/kg LY3015014 SC +Statin | 10.0 mg/kg LY3015014 IV | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/17
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 2/6 | 3/6 | 3/6 | 6/6 | 3/6 | 6/10 | 13/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.03 mg/kg LY3015014 IV (N=6) | 0.1 mg/kg LY3015014 IV (N=6) | 0.3 mg/kg LY3015014 IV (N=6) | 1.0 mg/kg LY3015014 IV (N=6) | 3.0 mg/kg LY3015014 IV (N=6) | 3.0 mg/kg LY3015014 SC (N=6) | 3.0 mg/kg LY3015014 SC +Statin (N=6) | 10.0 mg/kg LY3015014 IV (N=10) | Placebo (N=17)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram pr prolongation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased vibratory sense (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days